CLINICAL TRIAL: NCT01558388
Title: Randomised Control Trial of Probiotics Versus Placebo as Adjuvant to Oral Clindamycin Treatment for Bacterial Vaginosis During Pregnancy
Brief Title: Probiotic Versus Placebo as Adjuvant for Bacterial Vaginosis Treatment During Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Federico Prefumo, Consultant in Obstetrics and Gynaecology, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Spedali Civili 926
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal lactobacilli (Experimental)
  Interventions: Drug: Lactobacillus acidophilus
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus acidophilus — Lactobacillus acidophilus 500 million colony-forming units/tablets. One vaginal tablet daily for 10 days.
  Other Names: Pregyn-S
  Arms: Vaginal lactobacilli
Drug: Placebo — One vaginal tablet daily for 10 days.
  Arms: Placebo

SUMMARY:
Bacterial vaginosis is a common vaginal condition involving a reduction in the amount of Lactobacilli, the normal bacteria colonizing the vagina, and an overgrowth of pathogenic bacteria. The presence of bacterial vaginosis in pregnancy is associated with an increased risk of preterm delivery. After a course of antibiotic treatment, recurrence of bacterial vaginosis has been reported in 10-70% of cases. This study aims to verify if administration of vaginal Lactobacilli may reduce the occurrence rate after antibiotic treatment of bacterial vaginosis during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* gestational age 12-32 weeks
* diagnosis of bacterial vaginosis
* treatment of bacterial vaginosis with oral clindamycin 300 mg, twice-daily for 7 days

Exclusion Criteria:

* multiple pregnancy
* allergy to clindamycin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Vaginal lactobacillus recolonization | 3-5 weeks
Recurrence rate of bacterial vaginosis | 3-5 weeks

SECONDARY OUTCOMES:
Preterm delivery <37 weeks | within 43 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Luana Danti, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia; Andrea Lojacono, MD, Principal Investigator — Università degli Studi di Brescia
Locations (1):
- Ostetricia 1, Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Italy